CLINICAL TRIAL: NCT05989880
Title: Pilot Feasibility Trial of the SafeLM Supraglottic Airway
Brief Title: Pilot Feasibility Trial of the SafeLM Supraglottic Airway (SGA)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Lauren Nakazawa, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-23-0537
Record Dates: First submitted 2023-07-24; First posted 2023-08-14 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Anesthesia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- SafeLM as a supraglottic airway device with video capability (Experimental)
  Interventions: Device: SafeLM as a supraglottic airway device with video capability
- SafeLM as a supraglottic airway device without video capability (Experimental)
  Interventions: Device: SafeLM as a supraglottic airway device without video capability
- SafeLM as a conduit for intubation using an endotracheal tube with video capability (Experimental)
  Interventions: Device: SafeLM as a conduit for intubation using an endotracheal tube with video capability
- SafeLM as a conduit for intubation using a bougie with video capability (Experimental)
  Interventions: Device: SafeLM as a conduit for intubation using a bougie with video capability

INTERVENTIONS:
Device: SafeLM as a supraglottic airway device with video capability — The device will be inserted using the video capability and used as a primary airway device for the duration of the surgical procedure. Once the device is in place, the cuff will be inflated with the recommended volume of air to ensure an adequate seal around the laryngeal opening. The position of the device will be confirmed by observing the video image of the glottis on the monitor. The adequacy of ventilation and oxygenation will be assessed by monitoring the patient's end-tidal CO2, pulse oximetry, and clinical signs of effective ventilation. Leak and cuff pressure will be assessed. The device will be removed at the end of the surgical procedure or if there are any signs of device malfunction, airway obstruction, or inadequate ventilation.
  Arms: SafeLM as a supraglottic airway device with video capability
Device: SafeLM as a supraglottic airway device without video capability — The device will be blindly inserted without using the video capability and used as a primary airway device for the duration of the surgical procedure. Once the device is in place, the cuff will be inflated with the recommended volume of air to ensure an adequate seal around the laryngeal opening. The position of the device will be confirmed by observing the video image of the glottis on the monitor. The adequacy of ventilation and oxygenation will be assessed by monitoring the patient's end-tidal CO2, pulse oximetry, and clinical signs of effective ventilation. Leak and cuff pressure will be assessed. The video capability of the device will be used to assess the accuracy of placement after the fact. The device will be removed at the end of the surgical procedure or if there are any signs of device malfunction, airway obstruction, or inadequate ventilation.
  Arms: SafeLM as a supraglottic airway device without video capability
Device: SafeLM as a conduit for intubation using an endotracheal tube with video capability — The device will be inserted, and an endotracheal tube will be advanced through the device under direct visualization using the video capability of the device. Once the device is in place, the cuff will be inflated with the recommended volume of air to ensure an adequate seal around the laryngeal opening. The endotracheal tube will be introduced through the working channel of the SafeLM under direct visualization using the video capability of the device. The endotracheal tube will be advanced into the trachea, and the position will be confirmed by end-tidal carbon dioxide (EtCO2) detection and chest auscultation. The cuff of the endotracheal tube will be inflated, and mechanical ventilation will be resumed. The SafeLM device will be removed, and the position of the endotracheal tube will be confirmed once again.
  Arms: SafeLM as a conduit for intubation using an endotracheal tube with video capability
Device: SafeLM as a conduit for intubation using a bougie with video capability — The device will be inserted. Once the device is in place, the cuff will be inflated with the recommended volume of air to ensure an adequate seal around the laryngeal opening.The position of the device will be confirmed by observing the video image of the glottis on the monitor. The video camera on the SafeLM will be turned on to visualize the vocal cords.A standard airway bougie will be introduced through the working channel of the SafeLM under direct visualization using the video capability of the device.The SafeLM device will be removed, and an appropriately sized endotracheal tube will be advanced into the trachea. If a bougie is not able to be inserted into the tracheal under direct visualization, direct insertion of an endotracheal tube into the trachea will be attempted, followed by flexible scope intubation.
  Arms: SafeLM as a conduit for intubation using a bougie with video capability

SUMMARY:
The purpose of this study is to assess the feasibility of SafeLM as a primary airway device and as a conduit for intubation with and without the use of a bougie

ELIGIBILITY:
Inclusion Criteria:

* elective surgery requiring general anesthesia and airway management using a supraglottic airway device or endotracheal intubation

Exclusion Criteria:

* pregnancy
* known or suspected difficult airway management
* history of oropharyngeal or upper airway surgery
* known or suspected airway or respiratory pathology, such as significant obstructive sleep apnea or chronic obstructive pulmonary disease (COPD)
* BMI greater than 40 kg/m2
* unable to undergo intubation via the oral route
* known or suspected full stomach or other risk factors for aspiration
* contraindication for the use of neuromuscular blocking agents
* history of significant gastroesophageal reflux disease (GERD)
* Vulnerable populations (cognitively impaired persons, prisoners)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2025-10-02 (Estimated); Study Completion 2025-12-02 (Estimated)

PRIMARY OUTCOMES:
Intubation success rate | at the time of intubation
  This is assessed by the ability of the SafeLM to achieve adequate oxygenation and ventilation via the respective procedure once the airway device is in place.

SECONDARY OUTCOMES:
Number of insertion attempts required to achieve effective oxygenation and ventilation | at the time of intubation
Time to insertion | at the time of intubation
  This is measured by the time from opening the mouth to the time of end tidal CO2 on capnography
Subjective ease of insertion of the airway device | at the time of intubation
Safety of the SafeLM as an SGA | at the time of intubation
  This will be assessed by the number of adverse events such as airway obstruction, aspiration, and hypoxia.
Safety of the SafeLM as a conduit for intubation | at the time of intubation
  This will be assessed by the number of adverse events such as esophageal intubation, bronchial intubation, and hypoxia during the intubation process.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren M Nakazawa, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No